CLINICAL TRIAL: NCT02766959
Title: Bitter Taste and Allele-specific Expression of the Human TAS2R38 Gene
Brief Title: Allele-specific Expression of a Bitter Taste Receptor
Status: Completed | Type: Observational
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: University of Pennsylvania (Other); Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 823078
Record Dates: First submitted 2016-05-05; First posted 2016-05-10 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-01

CONDITIONS: Rhinosinusitis
Keywords: chronic rhinosinusitis; airway physiology; taste receptors; tas2r; epithelial biology; upper respiratory disease
MeSH Terms: conditions — Rhinosinusitis; Respiration Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In part one of the study, each subject will provide a saliva sample. DNA will be isolated, purified, and quantitated for alleles of TAS2R38, a bitter taste receptor gene. Based on the results of the genetic screen, 25 individuals with the heterozygous genotype will be invited to return for part two of the study. In part two of the study, subject will provide nasal epithelium and taste tissue in the form of fungiform papillae. One half of each set of tissue will be placed in saline on ice in preparation for cell culture and assessment of AHL-induced defensive responses, while the second half will be placed in RNA preservative for mRNA isolation.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PAV/PAV Tasters: Individuals homozygous for the taster allele of the TAS2R38 gene, PAV/PAV.
- AVI/PAV.: Individuals heterozygous for the taster allele of the TAS2R38 gene, AVI/PAV.
  Interventions: Other: Observational study
- AVI/AVI: Individuals homozygous for the non-taster allele of the TAS2R38 gene, AVI/AVI.

INTERVENTIONS:
Other: Observational study
  Groups: AVI/PAV.

SUMMARY:
This single-site, within-subject experimental basic research study is designed to analyze the hypothesis that allele-specific expression of the bitter taste receptor T2R38 in taste tissue of individuals heterozygous for the taste receptor gene TAS2R38 correlates with that in nasal epithelium, and is responsible for differences in acyl-homoserine lactone-induced respiratory defenses. Subjects will include 100 predominantly European adults without chronic rhinosinusitis who will be undergoing a sinonasal procedure for reconstructive purposes. All subjects will provide saliva samples for genotyping, from which 25 subjects heterozygous for TAS2R38 (AVI/PAV) will be identified. These individuals will be asked to complete a beverage frequency questionnaire and taste test prior to the procedure that will evaluate for a number of compounds, among them bitter ligands specific to T2R38. Their tongue will also be photographed to evaluate the anatomy of their fungiform papillae, the mushroom-like structures on the tongue which contain taste buds. Subjects will subsequently provide nasal epithelium and taste tissue, which will be processed to 1) evaluate for allele-specific expression of TAS2R38 mRNA in both the taste and nasal tissue, with the nasal tissue concurrently being cultured in an air-liquid interface system to 2) assess the AHL-induced respiratory defenses of ciliary beat frequency (CBF) and nitric oxide (NO) production. Should subjects require a subsequent sinonasal procedure for clinically-determined reasons, taste and nasal tissue will again be obtained and analyzed for TAS2R38 mRNA, allowing for 3) longitudinal evaluation of mRNA expression level.

DETAILED DESCRIPTION:
The Basic Biology of Bitter Taste. The perception of bitter taste is thought to have evolved as a mechanism to protect against the ingestion of toxic materials, and is the result of ligand-activation of one of more than 25 different bitter taste receptors, so-called T2Rs (1). These receptors are found on the tongue in what are called fungiform papillae, mushroom-like structures that contain taste buds with receptors responding to a variety of tastes including sweet, salty, sour, umami, and bitter. A prototypical example of one of these bitter ligands is phenylthiocarbamide (PTC), which actives the T2R38 receptor. While initially identified in type II taste cells, T2R38 is also expressed in nasal epithelium, where it participates in innate immune defense responses to invading bacteria (2-6).

TAS2R38: A Model System for Genotype-Phenotype Studies. Prior studies have identified two main forms of T2R38, active and inactive, which are characterized by three genetic variants in the TAS2R38 gene. These variants result in three amino acid changes, proline (P) to alanine (A) at position 49, alanine (A) to valine (V) at position 262, and valine (V) to isoleucine (I) at position 296 in the T2R38 receptor. Individuals who are homozygous for the active (PAV/PAV) form detect bitterness in compounds containing a thiourea (-N-C=S) moiety, including PTC, 6-n-propylthiouracil (PROP), and the plant compound goitrin, common in foods such as green vegetables (7-9). They also respond to acyl-homoserine lactones (AHLs), a class of compounds produced as signaling molecules by certain bacteria, triggering a rapid defense reaction consisting of increased ciliary beat frequency (CBF) to facilitate mucociliary clearance, and generation of nitric oxide (NO), a gas that can diffuse into the airway and kill bacteria (4). In contrast, those who are homozygous for all three variants (AVI/AVI) consume these compounds without perceiving them as bitter and do not appear to respond to AHLs (10). The frequency of both the active and inactive forms of TAS2R38 is at a near balance of 50:50 in many human racial groups, including Americans of European and African descent.

The Heterozygote Hypothesis. Interestingly, individuals heterozygous for the active form of the receptor (AVI/PAV) exhibit highly variable phenotypes, with some people very sensitive to bitter compounds, and others needing high concentrations to taste them at all (11). While the investigators know that taste papillae density plays at least some role in this variability

, our preliminary taste data suggest that the range of response is tied to how much mRNA is expressed from the active (PAV) form of the receptor, a concept called allele-specific expression (12). For example, this is the case when analyzing caffeine consumption, which strongly correlates with active mRNA expression (12). The investigators therefore hypothesize that the abundance of active TAS2R38 mRNA in heterozygous individuals also predicts the biologically significant change in magnitude of defensive responses in the presence of AHLs (13-15). The proposed study will determine whether this is in fact the case, and whether those people who have high mRNA abundance in taste tissue (fungiform papillae) also have correspondingly high abundance in nasal epithelium, or whether regulation is tissue-dependent. This will allow us to determine whether taste tests could provide a reliable representation of receptor function in other tissues and cell types. Should mRNA abundance prove to be a key factor, the investigators will determine whether high expressers sustain this expression over time.

Of note, a study performed by Dr. Reed and collaborators found that the population in Philadelphia contained 18% of individuals in the homozygous nontaster (AVI) group, 17% in the homozygous taster (PAV) group and 37% in the common heterozygous group (AVI/PAV) (16). The remaining 28% were distributed among ten other less common genotypes, which will not be analyzed in this study. Thus, as the majority of the population is heterozygous, a thorough understanding of their ability to fight infection is clinically important.

Clinical Significance. As one of the most common chronic conditions in the United States, chronic rhinosinusitis invokes a direct treatment cost of $3.5-5 billion annually. Its incidence is 146 per 1,000 and increasing (17). Our prior studies have shown that individuals with two copies of the active form of T2R38 have nasal epithelium that defends very effectively against certain bacteria, such as Pseudomonas aeruginosa, and are less likely to develop severe chronic rhinosinusitis requiring surgery, while those with two inactive forms cannot defend themselves as effectively, and are more likely to develop severe chronic rhinosinusitis requiring surgical intervention. Because the treatment of chronic rhinosinusitis involves multiple rounds of antibiotics and often surgical management through functional endoscopic sinus surgery (FESS), this research has significant implications for antibiotic stewardship, surgical morbidity and mortality, and health care expenditures.

ELIGIBILITY:
Inclusion Criteria:

* Key inclusion criteria include age 21-50 years
* English speaking, and plans to undergo a sinonasal procedure for reconstructive purposes or other reasons.

Exclusion Criteria:

* Key exclusion criteria include a history of chronic rhinosinusitis
* Plans to undergo a procedure for reasons other than reconstruction
* Oral disease
* Pregnancy, or any condition that would prevent psychophysical testing.
* Subjects showing signs of oral disease, including tongue lesions or xerostomia, would be excluded from tongue sampling, and therefore excluded from the study.
* Subjects will not be excluded because of economic status, gender, race or ethnicity.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: One hundred subjects will be tested for TAS2R38 genotype. Our typical subject population is approximately 82% of European descent and 35% female. All subjects will be recruited from those seen in the department of otorhinolaryngology's rhinology division and planning to undergo a sinonasal procedure for reconstructive purposes. The initial interview will occur in the clinic setting. From these 100 subjects, 25 who are heterozygous for TAS2R38 will be asked to perform a taste test, complete a beverage frequency questionnaire, have their tongue photographed, and provide nasal epithelium and taste tissue during their procedure. Key exclusion criteria include a history of chronic rhinosinusitis, oral disease, and any condition that would prevent them from completing the psychophysical testing.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
TAS2R38 genotype | Up to 1 month after enrollment.
  A participant's genotype will be identified on enrollment in the study, the results of which could take up to 1 month to be performed.
TAS2R38 mRNA expression levels measured by RT-qPCR | Approximately 6 weeks after subject enrollment
  Measured approximately 6 weeks after enrollment, based on the date of the participant's procedure.
Ciliary beat frequency | Approximately 6 weeks after subject enrollment
  Measured approximately 6 weeks after enrollment, based on the date of the participant's procedure.
Production of nitric oxide by a participant's nasal epithelium culture measured in fold change of 4,5-diaminofluorescence diacetate | Approximately 6 weeks after subject enrollment
  The production of nitric oxide (NO) by a patient's nasal epithelium culture will be measured approximately 6 weeks after enrollment, based on the date of his or her procedure. This will be measured by quantifying the fold change in fluorescence by using the NO-sensitive marker 4,5-diaminofluorescence diacetate (DAF-2).

SECONDARY OUTCOMES:
Bitter taste perception as measured by a visual analog scale | Approximately 6 weeks after subject enrollment
  Psychophysical bitter taste perception will be assessed by asking participants to taste a solution and rate its bitterness on a visual analog scale ranging from no intensity at all to extremely intense. This will be assessed at participant's post-procedure follow-up appointment, on average 6 weeks after enrollment.
Caffeine intake measured by number caffeinated beverages consumed per week (normalized to 1 cup = 180 mg caffeine) | Approximately 6 weeks after subject enrollment
  The scale will be normalized to 1 cup = 180 mg caffeine. This will be assessed at participant's post-procedure follow-up appointment, on average 6 weeks after enrollment.
Taste papillae density | Approximately 6 weeks after subject enrollment
  Papillae density will be assessed at participant's post-procedure follow-up appointment, on average 6 weeks after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle R. Reed, Ph.D., Principal Investigator — Monell Chemical Senses Center; Noam A. Cohen, M.D., Ph.D., Principal Investigator — Monell Chemical Senses Center, University of Pennsylvania
Locations (3):
- United States (3):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Monell Chemical Senses Center, Philadelphia, Pennsylvania
  - Philadelphia Veterans Affairs Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drewnowski A, Gomez-Carneros C. Bitter taste, phytonutrients, and the consumer: a review. Am J Clin Nutr. 2000 Dec;72(6):1424-35. doi: 10.1093/ajcn/72.6.1424. PMID 11101467
- [Background] Adler E, Hoon MA, Mueller KL, Chandrashekar J, Ryba NJ, Zuker CS. A novel family of mammalian taste receptors. Cell. 2000 Mar 17;100(6):693-702. doi: 10.1016/s0092-8674(00)80705-9. PMID 10761934
- [Background] Chandrashekar J, Mueller KL, Hoon MA, Adler E, Feng L, Guo W, Zuker CS, Ryba NJ. T2Rs function as bitter taste receptors. Cell. 2000 Mar 17;100(6):703-11. doi: 10.1016/s0092-8674(00)80706-0. PMID 10761935
- [Background] Lee RJ, Xiong G, Kofonow JM, Chen B, Lysenko A, Jiang P, Abraham V, Doghramji L, Adappa ND, Palmer JN, Kennedy DW, Beauchamp GK, Doulias PT, Ischiropoulos H, Kreindler JL, Reed DR, Cohen NA. T2R38 taste receptor polymorphisms underlie susceptibility to upper respiratory infection. J Clin Invest. 2012 Nov;122(11):4145-59. doi: 10.1172/JCI64240. Epub 2012 Oct 8. PMID 23041624
- [Background] Lee RJ, Kofonow JM, Rosen PL, Siebert AP, Chen B, Doghramji L, Xiong G, Adappa ND, Palmer JN, Kennedy DW, Kreindler JL, Margolskee RF, Cohen NA. Bitter and sweet taste receptors regulate human upper respiratory innate immunity. J Clin Invest. 2014 Mar;124(3):1393-405. doi: 10.1172/JCI72094. Epub 2014 Feb 17. PMID 24531552
- [Background] Tizzano M, Gulbransen BD, Vandenbeuch A, Clapp TR, Herman JP, Sibhatu HM, Churchill ME, Silver WL, Kinnamon SC, Finger TE. Nasal chemosensory cells use bitter taste signaling to detect irritants and bacterial signals. Proc Natl Acad Sci U S A. 2010 Feb 16;107(7):3210-5. doi: 10.1073/pnas.0911934107. Epub 2010 Jan 26. PMID 20133764
- [Background] Mueller KL, Hoon MA, Erlenbach I, Chandrashekar J, Zuker CS, Ryba NJ. The receptors and coding logic for bitter taste. Nature. 2005 Mar 10;434(7030):225-9. doi: 10.1038/nature03352. PMID 15759003
- [Background] Bufe B, Breslin PA, Kuhn C, Reed DR, Tharp CD, Slack JP, Kim UK, Drayna D, Meyerhof W. The molecular basis of individual differences in phenylthiocarbamide and propylthiouracil bitterness perception. Curr Biol. 2005 Feb 22;15(4):322-7. doi: 10.1016/j.cub.2005.01.047. PMID 15723792
- [Background] Wooding S, Bufe B, Grassi C, Howard MT, Stone AC, Vazquez M, Dunn DM, Meyerhof W, Weiss RB, Bamshad MJ. Independent evolution of bitter-taste sensitivity in humans and chimpanzees. Nature. 2006 Apr 13;440(7086):930-4. doi: 10.1038/nature04655. PMID 16612383
- [Background] Kim UK, Jorgenson E, Coon H, Leppert M, Risch N, Drayna D. Positional cloning of the human quantitative trait locus underlying taste sensitivity to phenylthiocarbamide. Science. 2003 Feb 21;299(5610):1221-5. doi: 10.1126/science.1080190. PMID 12595690
- [Background] Mennella JA, Pepino MY, Duke FF, Reed DR. Psychophysical dissection of genotype effects on human bitter perception. Chem Senses. 2011 Jan;36(2):161-7. doi: 10.1093/chemse/bjq106. Epub 2010 Oct 27. PMID 20980355
- [Background] Lipchock SV, Mennella JA, Spielman AI, Reed DR. Human bitter perception correlates with bitter receptor messenger RNA expression in taste cells. Am J Clin Nutr. 2013 Oct;98(4):1136-43. doi: 10.3945/ajcn.113.066688. Epub 2013 Sep 11. PMID 24025627
- [Background] Bartoshuk LM, Duffy VB, Miller IJ. PTC/PROP tasting: anatomy, psychophysics, and sex effects. Physiol Behav. 1994 Dec;56(6):1165-71. doi: 10.1016/0031-9384(94)90361-1. PMID 7878086
- [Background] Delwiche JF, Buletic Z, Breslin PA. Relationship of papillae number to bitter intensity of quinine and PROP within and between individuals. Physiol Behav. 2001 Oct;74(3):329-37. doi: 10.1016/s0031-9384(01)00568-6. PMID 11714496
- [Background] Melis M, Atzori E, Cabras S, Zonza A, Calo C, Muroni P, Nieddu M, Padiglia A, Sogos V, Tepper BJ, Tomassini Barbarossa I. The gustin (CA6) gene polymorphism, rs2274333 (A/G), as a mechanistic link between PROP tasting and fungiform taste papilla density and maintenance. PLoS One. 2013 Sep 9;8(9):e74151. doi: 10.1371/journal.pone.0074151. eCollection 2013. PMID 24040192
- [Background] Mennella JA, Pepino MY, Duke FF, Reed DR. Age modifies the genotype-phenotype relationship for the bitter receptor TAS2R38. BMC Genet. 2010 Jul 1;11:60. doi: 10.1186/1471-2156-11-60. PMID 20594349
- [Background] Pleis JR, Lucas JW. Summary health statistics for U.S. adults: National Health Interview Survey, 2007. Vital Health Stat 10. 2009 May;(240):1-159. PMID 19645319
- [Background] Suitor CJ, Gardner J, Willett WC. A comparison of food frequency and diet recall methods in studies of nutrient intake of low-income pregnant women. J Am Diet Assoc. 1989 Dec;89(12):1786-94. PMID 2592710
- [Background] Spielman AI, Pepino MY, Feldman R, Brand JG. Technique to collect fungiform (taste) papillae from human tongue. J Vis Exp. 2010 Sep 18;(42):2201. doi: 10.3791/2201. PMID 20972388